CLINICAL TRIAL: NCT03731871
Title: The Different Factors Involved in Fetal Maturity in Late Pregnancy
Brief Title: Parameters of Lung Maturity During Late Pregnancy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aljazeera Hospital (Other)
Collaborators: Kasr El Aini Hospital (Other); National Research Centre, Egypt (Other)
Responsible Party: Principal Investigator, Mahmoud Alalfy, Lecturer, Researcher , National Research centre and Specialist of Obstetrics and Gynecology in Aljazeerah hospital, Aljazeera Hospital
Other Study IDs: Lung
Record Dates: First submitted 2018-11-03; First posted 2018-11-06 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Pregnancy Related
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Ultrasonography — ultrasound to evaluate parameters of fetal maturity during pregnancy

SUMMARY:
- Lung maturity is one of the most important factors in perinatal medicine

DETAILED DESCRIPTION:
* Fetal development passes in many stages till fetal maturation occurs
* We are trying to line out fetal maturation

ELIGIBILITY:
Inclusion Criteria:

* pregnant ladies from 28 weeks till term

Exclusion Criteria:

* pregnant ladies before 28 weeks

Ages: 22 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant ladies
Study Population: pregnant ladies from 28 weeks till term
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-11-12 (Actual); Primary Completion 2020-07-15 (Estimated); Study Completion 2020-08-20 (Estimated)

PRIMARY OUTCOMES:
The number of fetuses who will be mature postnatally | within 2 weeks
  the neonates who willnot need incubators

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Alalfy, PhD, Study Chair — Algazeerah hospital -Location (Giza -Egypt ) and National Research centre egypt
Locations (1):
- Algazeerah and Kasralainy hospital, Giza, Egypt